CLINICAL TRIAL: NCT05784233
Title: Relevance and Salience During Attention Task
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 5R15EY030247-01A1 (NIH)
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: attention; visual search

STUDY DESIGN:
Intervention Model Description: All participants receive each level of task (easy singleton detection task, hard feature search task) and salient item presence (present, absent during search). Groups differ based on the likelihood of the salient item being the search target when present(0%-100%, in 25% increments).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 0% Relevance (Experimental): 0% chance of the salient item being the target during visual search task.
  Interventions: Behavioral: Relevance (Likelihood Salient Item is Target)
- 25% Relevance (Experimental): 25% chance of the salient item being the target during visual search task.
  Interventions: Behavioral: Relevance (Likelihood Salient Item is Target)
- 50% Relevance (Experimental): 50% chance of the salient item being the target during visual search task.
  Interventions: Behavioral: Relevance (Likelihood Salient Item is Target)
- 75% Relevance (Experimental): 75% chance of the salient item being the target during visual search task.
  Interventions: Behavioral: Relevance (Likelihood Salient Item is Target)
- 100% Relevance (Experimental): 100% chance of the salient item being the target during visual search task.
  Interventions: Behavioral: Relevance (Likelihood Salient Item is Target)

INTERVENTIONS:
Behavioral: Relevance (Likelihood Salient Item is Target) — The proportion of trials, when the salient visual item is present in the array, where the salient item is the search target.

SUMMARY:
In this line of research, the researchers are examining the influence of relevance of a salient item on task performance, depending on overall task set.

DETAILED DESCRIPTION:
When finding a target item during visual search (looking for a pencil), a salient item can capture attention (your phone flashing from a message). Typical attention studies only examine salient items when shown as distractor during search, to ensure any attention to the items are driven by salience alone. However, the impact of salience may interact with the relevance of the item for the search task (e.g. how likely the salient item is to be the target). Here, the researchers investigate these interactions in a basic science study when participants perform an easy task or a difficult search task.

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected to normal visual acuity, normal color vision

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Button Press Reaction Time | During Testing (single day)
  Speed to respond correctly to the target- after participant finds the target shape on a computer screen, they press a button to indicate what shape they see
Button Press Accuracy | During Testing (single day)
  Accuracy of responses to target item- the researchers will measure whether the participants presses the correct button which corresponds to the target shape presented on the computer screen or the incorrect button

CONTACTS AND LOCATIONS:
Locations (1):
- Lehigh University, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers plan to share anonymized subject data on Open Science Framework.
Supporting Information: Study Protocol
Time Frame: Upon publication.
Access Criteria: Open Science Framework, Internet access.